CLINICAL TRIAL: NCT05082129
Title: A Multicentre Pragmatic Clinical Investigation to Assess the Efficacy of TransiCap MRI Marker Device in Magnetic Resonance Imaging in Paediatric Constipation (MAGIC2)
Brief Title: Magnetic Resonance Imaging in Paediatric Constipation (MAGIC2)
Acronym: MAGIC2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to the impact of the COVID19 pandemic on MRI service provision, NHS hospitals were unable to provide the resources to conduct the study
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19GA038
Record Dates: First submitted 2021-03-24; First posted 2021-10-18 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2021-03

CONDITIONS: Constipation
Keywords: constipation; pediatric; transit
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention will consist of young patients with constipation presenting at secondary and tertiary care with intractable constipation. They will undergo the MRI gastrointestinal transit test (TransiCap). Their results will be shared with the patients after both MRI scans are preformed and results calculated. Their treatment selection will therefore be informed by the TransiCap results.
  Interventions: Device: TransiCap
- Control (Experimental): The control arm will consist of young patients with constipation presenting at secondary and tertiary care with intractable constipation. They will undergo the MRI gastrointestinal transit test (TransiCap). The patients will undergo 2 MRI scans but their results will be shared with the patients after 12 months has elapsed. They will receive standard care treatment not informed by the TransiCap results.
  Interventions: Device: TransiCap

INTERVENTIONS:
Device: TransiCap — The TransiCap device consists of small, completely inert mini-capsules that, once ingested, can be imaged inside the gastrointestinal tract using MRI, thereby creating a new MRI alternative to the radiopaque marker X-ray test to measure gut transit. The MRI mini- capsules are visualised in the gut using a single fat, water, in-phase and out-of-phase scan.

SUMMARY:
Constipation in children is a common problem. Managing these children is difficult, partly because they do not respond to laxatives and partly because their bowel problem cannot be defined. A "gut transit time" test can add information to help choose the best therapy but this is often not carried out because of the unsuitable radiation dose involved in the current methods such as X-ray. A new Magnetic Resonance Imaging (MRI) method to measure gut transit time using inert mini-capsules, the size of small pine nuts, has recently been developed and successfully trialled during a feasibility study.

This main multicentre study will trial the mini-capsules in 436 paediatric constipation patients.

DETAILED DESCRIPTION:
A fully powered, multi-centre, open label, pragmatic Randomised Controlled Trial (RCT) to test the use of the TransiCap MRI visible capsules to inform treatment selection and whether this leads to a change in rate of "treatment success" at 12 months after diagnosis.

Two study arms will include 436 young patients that present at secondary or tertiary care with constipation.

All participants will receive the TransiCap MRI Visible Capsules and the MRI scans at presentation, but only the participants in the intervention arm will have the results of their scan shared with the standard care team immediately. The intervention arm will therefore receive treatment which is informed by the TransiCap MRI transit time test. The participants in the control arm will instead receive standard care not informed by theTransiCap MRI visible capsules.

The results of the scans will be shared with the standard care team after the patient's follow up of 12 months is complete. All participants will receive the TransiCap MRI visible capsules and the MRI scans

ELIGIBILITY:
Inclusion Criteria:

Children aged 7 - 18 years old Able to give assent/consent or have a parent/carer able to give informed consent Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the clinical investigation.

Children diagnosed with clinical diagnosis of constipation

Exclusion Criteria:

The participant may not enter the clinical investigation if ANY of the following apply:

Female participants who are pregnant, lactating or planning pregnancy during the course of the clinical investigation. This will be self-reported.

Any history of gastrointestinal surgery that could affect gastrointestinal function, such as colectomy or small bowel resection.

Existing ACE procedure before the first MRI scan. Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury.

Inability to lie flat and relatively still for less than 5 minutes Poor understanding of English language Current diagnosis of COVID 19. The following disease or disorder; Bowel Stricture disease, Crohn's or any difficulty in swallowing (Dysphagia) Hirschsprung disease, congenital anorectal malformations, Paediatric Pseudo-obstruction syndrome

Currently using the following drugs influencing motility:

1. Opioid analgesics (tramadol, morphine, fentanyl, oxycodone, co-codamol and codydramoland)
2. Antispasmodic Buscopan (hyoscine butylbromide, also known as scopolamine butylbromide) Participants who have participated in another research clinical investigation involving an investigational product in the past 12 weeks.

4 or more bowel movements in one week and no episodes of bowel incontinence in one week (if these are reported in the participant's medical notes. Absence of this information should not warrant exclusion)

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-12 (Estimated); Primary Completion 2023-07-12 (Estimated); Study Completion 2023-07-12 (Estimated)

PRIMARY OUTCOMES:
Number of bowel movements | 12 months
  This outcome measure will be combined with the number of bowel incontinence episodes outcome to define the overall Treatment Success (yes/no) defined (from Rome IV criteria) as the patient achieving 3 or more bowel movements in one week and/or no episodes of bowel incontinence in one week at 12 months after the MRI study
Number of bowel incontinence episodes | 12 months
  This outcome measure will be combined with the number of bowel movements outcome to define the overall Treatment Success (yes/no) defined (from Rome IV criteria) as the patient achieving 3 or more bowel movements in one week and/or no episodes of bowel incontinence in one week at 12 months after the MRI study

SECONDARY OUTCOMES:
Whole gut transit time | Day 7
  Whole gut transit time (in hours) measured using the MRI visible mini-capsules
EQ-VAS | Day 7, 6 months and 12 months
  Visual analogue scale for health on the day
Adverse Events | 12 months
  Number of Adverse Events (AEs)
Serious Adverse Events | 12 months
  Number of Serious Adverse Events (SAEs)
Stool form | Day 7, 6 months and 12 months
  Bristol scale to measure stool form
Number of Mini-capsules swallowed | Day 4
  Number of Mini-capsules swallowed by the participants
Adverse Device Events | Day 7, 6 and 12 months
  Number of Adverse devise events recorded
AC-QoL | 12
  Adults (parents/carers) quality of life questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Hyman-Taylor, Study Director — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Upon completion external parties may request access to the data. Access to the data will be reviewed and approved by the data monitoring committee, funder and sponsor.
Supporting Information: Study Protocol
Time Frame: Upon completion of the study.
Access Criteria: to be determined